CLINICAL TRIAL: NCT04558502
Title: Effectiveness of Minocycline-Containing Bismuth Quadruple Therapy as First-Line Regimen for Helicobacter Pylori Eradication
Brief Title: Effectiveness of Minocycline-Containing Bismuth Quadruple Therapy for Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-584
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Helicobacter Pylori Eradication
Keywords: Helicobacter pylori; Eradication; minocycline; bismuth quadruple regimens
MeSH Terms: conditions — cyclopia sequence | interventions — Minocycline; Clarithromycin; Amoxicillin; Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- minocycline-based bismuth quadruple regimen for 14 days (Experimental): Esomeprazole 20 mg, minocycline 100 mg, amoxicillin 1000 mg, and colloidal bismuth pectin 200 mg twice daily for 14 days.
  Interventions: Drug: Minocycline hydrochloride capsule; Drug: Amoxicillin; Drug: colloidal bismuth pectin; Drug: esomeprazole
- clarithromycin-based bismuth quadruple regimen for 14 days (Active Comparator): Esomeprazole 20 mg,clarithromycin 500 mg, amoxicillin 1000 mg, and colloidal bismuth pectin 200 mg twice daily for 14 days.
  Interventions: Drug: Clarithromycin; Drug: Amoxicillin; Drug: colloidal bismuth pectin; Drug: esomeprazole
- minocycline-based bismuth quadruple regimen for 10 days (Experimental): Esomeprazole 20 mg, minocycline 100 mg, amoxicillin 1000 mg, and colloidal bismuth pectin 200 mg twice daily for 10 days.
  Interventions: Drug: Minocycline hydrochloride capsule; Drug: Amoxicillin; Drug: colloidal bismuth pectin; Drug: esomeprazole

INTERVENTIONS:
Drug: Minocycline hydrochloride capsule — Antibiotic for H. pylori eradication
  Other Names: Meiman
  Arms: minocycline-based bismuth quadruple regimen for 10 days; minocycline-based bismuth quadruple regimen for 14 days
Drug: Clarithromycin — Antibiotic for H. pylori eradication
  Other Names: Klacid
  Arms: clarithromycin-based bismuth quadruple regimen for 14 days
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: colloidal bismuth pectin — Gastric mucosal protective drug with anti-H. pylori effect
Drug: esomeprazole — Proton pump inhibitor

SUMMARY:
Although,bismuth-containing quadruple therapy has been highly recommended as first-line treatment regimen for H.pylori infection,it also has its problems and limitations in China.The primary resistance rates of metronidazole,clarithromycin and levofloxacin are all high in China.Besides that,tetracycline cannot be obtained and its complicated administration (four times daily) easily reduce patient compliance. In this study, we proposed to evaluate the eradication rate, safety, and compliance of a minocycline-based bismuth quadruple regimen.

DETAILED DESCRIPTION:
A total of 339 H. pylori-infected, treatment-naive patients will be enrolled in this randomized controlled clinical trial. Patients will be randomly allocated into 3 groups: Esomeprazole 20 mg, clarithromycin 500 mg, amoxicillin 1000 mg, and colloidal bismuth pectin 200 mg twice daily for 14 days; Esomeprazole 20 mg, minocycline 100 mg, amoxicillin 1000 mg, and colloidal bismuth pectin 200 mg twice daily for 14 days; Esomeprazole 20 mg, minocycline 100 mg, amoxicillin 1000 mg, and colloidal bismuth pectin 200 mg twice daily for 10 days. Eradication rates will be assessed 4-12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* H.pylori-positive outpatients with endoscopically proven chronic gastritis
* H. pylori (+) determined by either the 14C-or 13C-urea breath test or the gastric mucosal tissue rapid urease test and pathological section staining
* Treatment-naive patients for eradication of H.pylori infection
* Fully informed and agreed to participate in this study

Exclusion Criteria:

* Age <18 years or >70 years
* Allergy to any of the study drugs
* Use of any drug that could influence the study results 4 weeks before the study,such as antibiotics,bismuth agent,PPI or H2 receptor antagonist (H2RA)
* Previous gastric or esophageal surgery
* Patients with malignancy or severe comorbidity
* Pregnancy,lactation or alcohol abuse
* Patients with poor treatment compliance or could not express themselves correctly
* Participation in other clinical studies recently (within 3 months of enrollment in this clinical study)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Estimated)
Dates: Start 2022-01-05 (Estimated); Primary Completion 2022-06-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 4-12 weeks after treatment
  Helicobacter pylori eradication of minocycline-containing bismuth quadruple therapy

SECONDARY OUTCOMES:
incidence of adverse effects | 3-7 days after treatment
  incidence of adverse effects of minocycline-containing bismuth quadruple therapy

CONTACTS AND LOCATIONS:
Overall Officials: Qin Du, master, Principal Investigator — 2nd Affiliated Hospital,School of Medicine,Zhejiang University,China

IPD SHARING:
Plan to Share IPD: No